CLINICAL TRIAL: NCT00735072
Title: Maraviroc as an Immunomodulatory Drug for Antiretroviral-treated HIV Infected Patients Exhibiting Immunologic Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry); amfAR, The Foundation for AIDS Research (Other); Stanford University (Other); Case Western Reserve University (Other); Rush University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA9001DE
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Results first posted 2012-07-18 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infection
Keywords: HIV infection; T cell activation; Antiretroviral Therapy; CCR5; Maraviroc
MeSH Terms: conditions — HIV Infections | interventions — Maraviroc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maraviroc (Experimental): Maraviroc (dose based on current medications in regimen: 150mg orally (PO) twice daily (BID) for those on a protease inhibitor-based regimen other than Tipranavir; 600mg PO BID for efavirenz-containing regimens; or 300 mg PO BID for all other regimens).
  Interventions: Drug: Maraviroc
- Placebo (Placebo Comparator): Placebo (dose based on current medications in regimen: 150mg PO BID for those on a protease inhibitor-based regimen other than Tipranavir; 600mg PO BID for efavirenz-containing regimens; or 300 mg PO BID for all other regimens).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Dose based on current medications in regimen: 150mg PO BID for those on a protease inhibitor-based regimen other than Tipranavir; 600mg PO BID for efavirenz-containing regimens; or 300 mg PO BID for all other regimens.
  Other Names: Placebo for Maraviroc
  Arms: Placebo
Drug: Maraviroc — Dose based on current medications in regimen: 150mg orally (PO) twice daily (BID) for those on a protease inhibitor-based regimen other than Tipranavir; 600mg PO BID for efavirenz-containing regimens; or 300 mg PO BID for all other regimens.
  Other Names: Selzentry
  Arms: Maraviroc

SUMMARY:
Many people with HIV fail to regain normal CD4 counts despite effectively suppressing HIV replication with medications. Blocking the "co-receptor" for HIV might decrease inflammation of the immune system, potentially providing an immune benefit. The goal of the current trial is to determine whether adding maraviroc, a new CCR5 "co-receptor" blocker, decreases inflammation, providing an immune benefit for patients with low CD4 counts despite undetectable viral loads on HIV medications.

In this study, HIV-infected patients who are receiving antiretroviral therapy for HIV will receive either maraviroc or a placebo (sugar pill) each day for 24 weeks. After 24 weeks, the study medication will be stopped and all subjects will be followed for 12 more weeks. Blood tests measuring the extent of inflammation, low-level viremia, and immune function will be measured throughout the trial and compared between treatment arms.

DETAILED DESCRIPTION:
Our primary hypothesis is that CCR5 inhibitors may have protective immunomodulatory effects independent of their impact on HIV replication. Specifically, we predict that maraviroc will reduce the persistent T cell activation that prevents normal immune reconstitution during HAART-mediated viral suppression. This hypothesis will be tested in the context of a placebo controlled pilot study assessing the impact of maraviroc in antiretroviral-treated patients with a CD4+ T cell count less than 350 cells/mm3. In order to address the immunologic activity of this drug independent of plasma HIV RNA levels, we will study individuals who have undetectable viral loads (< 75 copies RNA/mL). Subjects will be randomized to maraviroc for 24 weeks or matching placebo for 24 weeks, followed by a 12 week washout period. We will use as our primary endpoint the proportion of CD8+ T cells that co-expresses CD38 and HLA-DR, as these outcomes have been well validated in prior studies. The primary outcome will be change in the percentage of activated CD8+ T cells at week 24. Change in CD4+ T cell counts, HIV RNA levels (using ultra-sensitive techniques), and other more experimental immunologic measurements will be assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test.
2. Stable antiretroviral therapy for at least 12 months
3. Screening CD4+ T cell count below 350 cells/mm3
4. All available CD4+ T cell counts in the last year and at screening < 350 cells/mm3
5. Screening plasma HIV RNA levels below level of detection (< 50 copies RNA/mL using Roche Amplicor or < 75 copies/mL using Bayer bDNA)
6. All available plasma HIV RNA levels within past year below the level of detection. Isolated values that are detectable but < 500 copies will be allowed as long as the plasma HIV RNA levels before and after this time point are undetectable.
7. > 90% adherence to therapy within the preceding 30 days, as determined by self-report.
8. Both male and female subjects are eligible. Females of childbearing potential must have a negative serum pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.
9. Ability and willingness of subject or legal guardian/representative to provide informed consent

Exclusion Criteria:

1. Increase in CD4 count of > 100 cells/mm3 in past year.
2. Patients who are intending to modify antiretroviral therapy in the next 24 weeks for any reason.
3. Serious illness requiring hospitalization or parental antibiotics within preceding 3 months.
4. Concurrent treatment with immunomodulatory drugs, or exposure to any immunomodulatory drug in past 16 weeks.
5. HBVsAg+ or active hepatitis C or hepatitis B which will require treatment in the subsequent 24 weeks.
6. Prior exposure to CCR5 inhibitors
7. Screening absolute neutrophil count <1,000 cells/mm3, platelet count <50,000 cells/mm3, hemoglobin < 8mg/dL, estimated creatinine clearance <40 mL/minute.
8. Pregnant or breastfeeding women
9. Use of both Tenofovir and Didanosine in current antiretroviral therapy regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Hunt, MD, Principal Investigator — University of California, San Francisco; Steven G Deeks, MD, Principal Investigator — University of California, San Francisco; Nancy Shulman, MD, Principal Investigator — Stanford University; Robert Shafer, MD, Principal Investigator — Stanford University; Michael Lederman, MD, Principal Investigator — Case Western Reserve University; Toyin Adeyemi, MD, Principal Investigator — Rush University
Locations (4):
- United States (4):
  - University of California San Francisco - San Francisco General Hospital, San Francisco, California
  - Stanford University, Stanford, California
  - Rush University - Stroger Hospital of Cook County, Chicago, Illinois
  - Case Western Reserve University, Cleveland, Ohio

REFERENCES:
- [Derived] Hunt PW, Shulman NS, Hayes TL, Dahl V, Somsouk M, Funderburg NT, McLaughlin B, Landay AL, Adeyemi O, Gilman LE, Clagett B, Rodriguez B, Martin JN, Schacker TW, Shacklett BL, Palmer S, Lederman MM, Deeks SG. The immunologic effects of maraviroc intensification in treated HIV-infected individuals with incomplete CD4+ T-cell recovery: a randomized trial. Blood. 2013 Jun 6;121(23):4635-46. doi: 10.1182/blood-2012-06-436345. Epub 2013 Apr 15. PMID 23589670

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the HIV clinics at San Francisco General Hospital, Stanford University, Case Western Reserve University, and Rush University/CORE Center between September, 2008, and December, 2009.
Pre-assignment Details: All 45 enrolled patients were assigned to study intervention. We over-enrolled by 3 subjects given 2 premature treatment discontinuations and one subject with unavailable baseline peripheral blood mononuclear cell (PBMC) samples available for analysis.
Groups:
- Maraviroc: Maraviroc (dose based on current medications in regimen: 150mg PO BID for those on a protease inhibitor-based regimen other than Tipranavir; 600mg PO BID for efavirenz-containing regimens; or 300 mg PO BID for all other regimens).
Period: Overall Study
Arm/Group | Maraviroc | Placebo
Started | 23 | 22
Completed | 22 | 21
Not Completed | 1 | 1
Not completed — interrupted study med during ARV change | 1 | 0
Not completed — Subject interrupted ARVs (non-adherence) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc | Placebo | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 44
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (8) | 50 (10) | 50 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 23 | 20 | 43
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Week 24 Change in Percentage of CD8+ T Cells That Co-express CD38 and HLA DR (Week 24 %CD38+HLA-DR+ CD8+ T Cells Minus Baseline %CD38+HLA-DR+ CD8+ T Cells)
Time Frame: Baseline and Week 24
Measure: Median (Inter-Quartile Range); unit: %CD38+ HLA-DR+ CD8+ T cells
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 23 | 22
%CD38+ HLA-DR+ CD8+ T cells | 2.2 [-0.6 to 4.1] | -0.7 [-3.5 to 0.6]
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; Null hypothesis: there will be no difference in the week 24 change in %activated CD8+ T cells between arms. Assuming a standard deviation as high as 3.5% and a Type I error of 5%, with 21 subjects in each treatment arm we would have 80% statistical power to detect a mean 3 percentage-point difference in the percent of activated CD8+ T cells between the active drug and placebo groups; Test type: Superiority or Other; p = 0.014, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in CD4+ T Cell Count
Time Frame: Baseline and Week 24
Measure: Mean (95% Confidence Interval); unit: cells/mm^3 over 24 weeks
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 22 | 21
cells/mm^3 over 24 weeks | 17 [7 to 28] | 17 [7 to 27]
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; Test type: Other; p = 0.97, Mixed Models Analysis

3. Secondary Outcome: Change in Ultra-sensitive Plasma HIV RNA Level (Single Copy/ml Assay)
Time Frame: Baseline and Week 24
Population: Data available only on the 35 participants with at least 7 mL of plasma available as reported here.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 18 | 17
percent change from baseline | -52 [-68 to -22] | -48 [-72 to -4]
Statistical Analysis 1: Comparison: Maraviroc vs Placebo; Test type: Other; p = 0.33, Mixed Models Analysis

4. Secondary Outcome: Change in Brachial Artery Flow-mediated Dilatation (UCSF Site Only)
Time Frame: Baseline and Week 24
Population: These data were collected from participants enrolled at the UCSF site only, as reported here.
Measure: Mean (95% Confidence Interval); unit: percent change from baseline
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 10 | 9
percent change from baseline | 1.0 [-0.5 to 2.5] | 0.3 [-1.1 to 1.8]

5. Secondary Outcome: Change in Gut-associated Lymphoid Tissue HIV RNA Level (UCSF Site Only)
Time Frame: Baseline and Week 24
Population: These data were collected from participants enrolled at the UCSF site only, as reported here.
Measure: Median (Inter-Quartile Range); unit: percent change from baseline
Arm/Group | Maraviroc | Placebo
Number analyzed (Participants) | 6 | 6
percent change from baseline | -11 [-26 to 23] | -3 [-43 to 91]

ADVERSE EVENTS:
Time Frame: 36 weeks
Arm/Group | Maraviroc | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 4/23 | 2/22
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Maraviroc (N=23) | Placebo (N=22)
Indirect Hyperbilirubinemia (on atazanavir-based ART) (Hepatobiliary disorders) | 2 | 1 — All cases were comparable to baseline values and all were on atazanavir-based regimens. None required treatment change during the trial.
Prolonged Fever (Infections and infestations) | 1 | 0 — Unexplained fever for 2 weeks without identifiable cause, resolved in absence of any specific therapy and subject had continued study medication without recurrence.
Triglyceride Elevation (Metabolism and nutrition disorders) | 1 | 0 — Grade 3 trygliceride elevation noted, comparable to recent values prior to enrollment and resolved to baseline values without change in therapy.
HBV flare, transaminitis (Hepatobiliary disorders) | 0 | 1 — Subject stopped all ARVs and study medications due to a lapse in insurance coverage (and didnt notify physician or study team). Had a recurrence of HBV viremia with transaminitis (after discontinuing study medication), resolved after restarting ART.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No